CLINICAL TRIAL: NCT01608984
Title: Effects of Remote Ischemic PreConditioning in Off-pump Versus On-pump Coronary
Brief Title: Effects of Remote Ischemic PreConditioning in Off-pump Versus On-pump Coronary Artery Bypass Grafting(RIPCON)
Acronym: RIPCON
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: University Hospital, Essen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RIPCON-12
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Myocardial Injury
Keywords: remote ischemic preconditioning; coronary artery bypass grafting; myocardial injury
MeSH Terms: interventions — Isoflurane; Sufentanil; Coronary Artery Bypass

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- RIPC-CABG (Active Comparator): Remote ischemic preconditioning (RIPC) protocol before coronary artery bypass surgery with blood cardioplegia for cardiac arrest (CABG) consists of 3 cycles of 5 minutes left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 minutes of reperfusion after induction of anesthesia before coronary artery bypass surgery. For myocardial molecular analyses, left ventricular biopsies are taken before induction of cardioplegic cardiac arrest and 5 to 10 Minutes after aortic unclamping during reperfusion of the myocardium. Blood samples are taken up to 72 hours postoperatively.
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- Control-CABG (Placebo Comparator): Control group: Coronary artery bypass grafting without RIPC protocol
  Interventions: Procedure: Coronary artery bypass grafting (CABG) without remote ischemic preconditioning protocol
- RIPC-OPCAB (Active Comparator): Remote ischemic preconditioning (RIPC) protocol before Off-pump coronary artery bypass surgery (OPCAB) consists of 3 cycles of 5 minutes left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 minutes of reperfusion after induction of anesthesia before coronary artery bypass surgery. For myocardial molecular analyses, left ventricular biopsies are taken before first coronary artery incision and 5 to 10 Minutes after completion of the coronary anastomoses. Blood samples are taken up to 72 hours postoperatively.
  Interventions: Procedure: Remote ischemic preconditioning (RIPC)
- Control-OPCAB (Placebo Comparator): Control group: Off-pump Coronary artery bypass surgery without RIPC protocol
  Interventions: Procedure: Off-pump Coronary artery bypass surgery without remote ischemic preconditioning

INTERVENTIONS:
Procedure: Remote ischemic preconditioning (RIPC) — 3 cycles of 5 min left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 min reperfusion.
  The applied anesthesia protocol avoids the use of propofol. Drugs: isoflurane+sufentanil anesthesia Anaesthesia is maintained by inhaled isoflurane in concentrations 0.7-0.8 % end-tidal with additional sufentanil injected during surgery, as required. In the CABG-arms, during extracorporal circulation patients receive isoflurane via a vaporizer incorporated in the extracorporeal gas supply in the same concentrations.
  Other Names: RIPC: remote ischemic preconditioning; CABG: coronary artery bypass grafting; OPCAB: Off-pump coronary artery bypass surgery; Isoflurane: 2-chloro-2-(difluoromethoxy)-1,1,1-trifluoro-ethane, Forane; Sufentanil, Sufenta, (R-30730)
  Arms: RIPC-CABG; RIPC-OPCAB
Procedure: Coronary artery bypass grafting (CABG) without remote ischemic preconditioning protocol — The applied anesthesia protocol avoids the use of propofol. Drugs: isoflurane+sufentanil anesthesia Anaesthesia is maintained by inhaled isoflurane in concentrations 0.7-0.8 % end-tidal with additional sufentanil injected during surgery, as required. During extracorporal circulation patients receive isoflurane via a vaporizer incorporated in the extracorporeal gas supply in the same concentrations.
  Arms: Control-CABG
Procedure: Off-pump Coronary artery bypass surgery without remote ischemic preconditioning — The applied anesthesia protocol avoids the use of propofol. Drugs: isoflurane+sufentanil anesthesia Anaesthesia is maintained by inhaled isoflurane in concentrations 0.7-0.8 % end-tidal with additional sufentanil injected during surgery, as required.
  Arms: Control-OPCAB

SUMMARY:
Purpose Remote ischemic preconditioning (RIPC) with transient upper limb ischemia reduces myocardial injury in patients undergoing On-pump coronary artery bypass (CABG) surgery with cross-clamp fibrillation or blood cardioplegia for myocardial protection. The molecular mechanisms leading to these effects are yet not fully understood. The purpose of the present study is to validate previous studies and gather further evidence for RIPC during CABG with blood cardioplegia, furthermore to determine, whether or not RIPC is still operative during Off-pump coronary artery bypass surgery (OPCAB), finally to elucidate intra-cellular mechanisms involved in myocardial protection by RIPC and their possible systemic mediators.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) protocol before CABG (study arm A) or OPCAB (study arm B) consists of 3 cycles of 5 minutes left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 minutes of reperfusion after induction of anesthesia before coronary artery bypass surgery. For myocardial molecular analyses, left ventricular biopsies are taken before induction of cardioplegic cardiac arrest (A) or first coronary incision (B), and 5 to 10 minutes after aortic unclamping during reperfusion of the myocardium (A) or 5 to 10 minutes after the completion of the last anastomosis (B). Blood samples are taken prior to RIPC and during the first three postoperative days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed triple vessel coronary artery disease
* Indication for surgical coronary revascularisation
* Written informed consent
* Age ≥ 18 years

Exclusion Criteria:

* Age > 80 years
* Instable angina/acute coronary syndrome
* Emergency surgery
* Recent myocardial infarction within 7 days prior to surgery
* Recent major infection/sepsis within 7 days prior to surgery
* Significant hepatic, renal oder pulmonary disease
* Other concomitant surgical procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative extent of myocardial injury as measured by cardiac troponin T serum release over 72 hours after coronary bypass surgery and its area under the curve (AUC). | 72 hours postoperatively after CABG surgery

SECONDARY OUTCOMES:
All-cause mortality | 30 days and 1 year after coronary bypass surgery
Major adverse cardiac and cerebrovascular events (MACCE) | 30 days and 1 year after coronary bypass surgery
Myocardial infarction | 30 days and 1 year after coronary bypass surgery
Renal function | 30 days and 1 year after coronary bypass surgery
circulating microparticles after coronary bypass surgery | perioperatively, 3 months and 1 year after coronary bypass surgery

CONTACTS AND LOCATIONS:
Overall Officials: Payam Akhyari, MD, Principal Investigator — Dept. of Cardiovascular Surgery, University Hospital, Heinrich Heine University, Duesseldorf, Germany; Alexander Albert, MD, Principal Investigator — Dept. of Cardiovascular Surgery, University Hospital, Heinrich Heine University, Duesseldorf, Germany; Artur Lichtenberg, MD, Principal Investigator — Dept. of Cardiovascular Surgery, University Hospital, Heinrich Heine University, Duesseldorf, Germany; Gerd Heusch, MD, PhD, Principal Investigator — nst. of Pathophysiology, University Duisburg-Essen, University Hospital Essen, Essen, Germany
Locations (1):
- Dept. Cardiovascular Surgery, University Hospital, Heinrich Heine University, Düsseldorf, Germany

REFERENCES:
- [Background] Hausenloy DJ, Erik Botker H, Condorelli G, Ferdinandy P, Garcia-Dorado D, Heusch G, Lecour S, van Laake LW, Madonna R, Ruiz-Meana M, Schulz R, Sluijter JP, Yellon DM, Ovize M. Translating cardioprotection for patient benefit: position paper from the Working Group of Cellular Biology of the Heart of the European Society of Cardiology. Cardiovasc Res. 2013 Apr 1;98(1):7-27. doi: 10.1093/cvr/cvt004. Epub 2013 Jan 19. PMID 23334258
- [Background] Heusch G, Musiolik J, Kottenberg E, Peters J, Jakob H, Thielmann M. STAT5 activation and cardioprotection by remote ischemic preconditioning in humans: short communication. Circ Res. 2012 Jan 6;110(1):111-5. doi: 10.1161/CIRCRESAHA.111.259556. Epub 2011 Nov 23. PMID 22116817